CLINICAL TRIAL: NCT02094521
Title: Evaluation of Optimal Dosing Conditions for GLP-1 Analogue NNC0113-0987 When Administered Orally in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9926-4047; 2012-003855-13 (EudraCT Number); U1111-1133-7097 (Other: WHO)
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NNC0113-0987 (Experimental)
  Interventions: Drug: NNC0113-0987

INTERVENTIONS:
Drug: NNC0113-0987 — For oral administration. All subjects will be treated for 10 consecutive days with five days on 5 mg NNC0113-0987 followed by five days on 10 mg NNC0113-0987. Dose escalation is chosen to increase gastrointestinal tolerability.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to evaluate the optimal dosing conditions for GLP-1 analogue NNC0113-0987 when administered orally in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 between 55 years (both inclusive) at the time of signing informed consent
* Good general health based on medical history, physical examination, and results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator
* Body mass index (BMI) between 18.5 and 29.9 kg/m^2 (both inclusive)

Exclusion Criteria:

* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular,respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Blood pressure above 140 mmHg systolic and/or above 90 mmHg diastolic or pulse above 90 beats per minute at the screening visit
* Smoking more than 5 cigarettes or the equivalent per day (including use of nicotine substitute products)
* History of significant drug abuse, or a positive drug test at the screening visit
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding the screening visit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area under the NNC0113-0987 plasma concentration time curve | From time 0 to 24 hours after the 10th dosing

SECONDARY OUTCOMES:
Maximum observed NNC0113-0987 plasma concentration | 0 to 24 hours after the 10th dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Harrow, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com